CLINICAL TRIAL: NCT05725616
Title: Effectiveness of the Anatomical Snuff Box Approach for Coronary Angiography: Comparative Non-inferiority Study With the Radial Arterial Approach to the Wrist
Brief Title: Effectiveness of the Anatomical Snuff Box Approach for Coronary Angiography
Acronym: COROTAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A01928-35
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Coronary Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snuff box puncture (Experimental): Puncture of the radial artery at of the anatomical snuff box or on the back of the hand during coronary angiography
  Interventions: Procedure: Coronary angiography
- Wrist puncture (Active Comparator): Puncture of the radial artery at the level of the base of the wrist during coronary angiography
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Coronary angiography — Snuff Box Approach or radial Arterial Approach at wrist for coronary angiography.

SUMMARY:
The main objective of the study is to assess whether the distal radial arterial approach (snuff box or back of the hand) is not inferior to the radial arterial approach at the wrist, in the management of coronary angiography for diagnostic purposes

DETAILED DESCRIPTION:
Coronary angiography is the reference examination for anatomical exploration coronary arteries to determine the presence or absence of a predominantly obstructive coronary disease.

Historically, the femoral approach was the most common approach used in interventional cardiology. The radial approach to the forearm presents multiple advantages over the femoral route, and it became the gold standard approach to coronary angiography and intervention percutaneous coronary. Although uncommon, vascular complications related to the radial pathway exist.

This is why a more distal radial approach, above the long tendon extensor of the thumb (at the level of the anatomical snuff box) or downstream (at the back of the hand) was suggested more than 10 years ago. This pathway is now an advantageous alternative to the radial approach of first intention, both for the patient and for the practitioner.

The two procedures are common today but few studies have been developed to compare the two approaches. Therefore, the main objective of the study is to assess whether the distal radial arterial approach (snuff box or back of the hand) is not inferior to the radial arterial approach at the wrist, in the management of coronary angiography for diagnostic purposes

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 and over
* Patient having a diagnostic coronary angiography programmed by radial route.
* Patient with a radial pulse at the anatomical snuff box and at the wrist noticeable

Exclusion Criteria:

* Patient requiring emergency coronary angiography or having an acute coronary syndrome
* Patient with severe arteriopathy of the supra-aortic trunks
* Patient with a history of coronary bypass surgery
* Tall patients (>1.90m)
* Patient allergic to xylocaine
* Patient presenting a contraindication to the realization of a coronary angiography:

terminal IRC, pregnancy, severe sepsis....

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Success rate of coronary angiography without changing puncture route. | 1 day
  The primary endpoint is the success rate of coronary angiography without changing puncture route.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiologie Tonkin, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No